CLINICAL TRIAL: NCT04164524
Title: Professor and HOD Department of Surgery DIMC
Brief Title: Frequency of Surgical Site Infection in Abdominal Hernia With Gentamycin Spray on Mesh Versus no Spray
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shahida Parveen Afridi, Professor of Surgery, Dow University of Health Sciences
Other Study IDs: 1883
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Wound With Foreign Body (With or Without Infection)
Keywords: SSI; Wound infection
MeSH Terms: conditions — Wound Infection | interventions — Gentamicins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group; A: Open technique Hernioplasty for abdominal hernia in which 160 mg Gentamycin spray applied over the mesh
  Interventions: Drug: Gentamycin
- Group; B: Open technique Hernioplasty for abdominal hernia in which no Gentamycin spray applied over the mesh

INTERVENTIONS:
Drug: Gentamycin — Gentamycin 160 mg spray applied over the mesh
  Groups: Group; A

SUMMARY:
Patient diagnosed with Para umbilical hernia, umbilical hernia, epigastric will be selected for the study. Sampling technique will be systematic with every 2nd patient being exposed to Gentamycin spray during mesh repair. . Each procedure took 90 to 120 minutes approximately. All patients underwent open abdominal hernioplasty operated on elective list. After placing onlay polypropylene mesh fixed with 2-0 prolene and gentamicin 160 mg injection will be sprayed over the secured mesh. Close active suction drain will be placed in subcutaneous space. Finally we will close the skin with Prolene 2-0 with vertical mattress suture or stapler.

DETAILED DESCRIPTION:
Patients and methods:

The study will be conducted at Dow University Hospital Karachi, Ojha Campusa. The subjects included were elective patients operated for abdominal hernias. Sample size calculated for a larger study with 50% frequency, and 99% confidence levels, using Openepi was found to be 664. According to Connelly*, the sample size of pilot study should be 10% of the sample size of a larger pilot study. As it is a pilot study, the sample size for this study was found to be 66.

We will take the informed consent before including the patient in the study. Inclusion criteria Following hernia operated on elective list

* Para umbilical hernia
* Umbilical hernia
* Epigastric hernia

Exclusion criteria

* All above hernia operated in emergency
* Inguinal hernia

Sampling technique will be systematic with every 2nd patient being exposed to Gentamycin spray during mesh repair. . Each procedure took 90 to 120 minutes approximately. All patients underwent open abdominal hernioplasty operated on elective list. After placing onlay polypropylene mesh, fixed with 2-0 prolene and gentamicin 160 mg injection will be sprayed over the secured mesh. Close active suction drain will be placed in subcutaneous space. Finally skin will be close with Prolene 2-0 with vertical mattress suture or stapler. All patients discharge on a day care basis with follow-ups in the OPD Out patient Department for any post-operative SSI Surgical site infection for a period of two weeks. Drains will be remove once no or less than 20 ml serosanguinous/ serous discharge in 24 hours.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery; Para umbilical hernia, umbilical and epigastric hernia,

Exclusion Criteria:

Emergency Admission incissional hernia inguinal hernia

-

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Two group Study population selected from Out patient Department for elective Surgery
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Wound infection | two weeks
  SSI Surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Shahida Parveen Afridi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Through research paper
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 month
Access Criteria: email